CLINICAL TRIAL: NCT06652373
Title: Evaluation of The Effectiveness of Perinatal Bereavement Counseling Training for Midwives
Brief Title: Perinatal Bereavement Counseling Training for Midwives
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayşe İrem Gökçek, PhD student in midwifery, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IUC-EBE-AIG-01
Record Dates: First submitted 2024-09-12; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Still Births; Bereavement; Perinatal Care; Perinatal Mental Health
Keywords: Bereavement; Hospice Care; Research Design; Midwifery; Pregnancy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): perinatal grief counselling training for midwives will be given to the experimental group.
  Interventions: Behavioral: Behavioural change through education
- Standard of care (No Intervention): The training will not be given to the control group during the study.

INTERVENTIONS:
Behavioral: Behavioural change through education — The content of the perinatal grief counselling training to be used in the study will be created in 8 modules and will be applied to midwives. The planned perinatal grief counselling training for midwives will be carried out online and it is aimed that midwives gain perinatal grief counselling skills and competence and increase their competence to cope with the problems they may encounter in the counselling process.
  Arms: Education

SUMMARY:
Perinatal bereavement is a condition that can lead to serious psychological problems for parents and their families. Bereaved women are at high risk of mental health problems (e.g. anxiety, post-traumatic stress disorder and depression). They may also blame themselves and their bodies for the loss and feel inadequate. Inadequate support from their environment in this process may lead them to experience social isolation. Research highlights the impact of caring for bereaved parents on health professionals, and that inadequate training can have a negative impact. In this context, there is a need for well-structured and tailored training programmes that focus on the specific needs and skills required to provide appropriate bereavement care to parents experiencing pregnancy loss and perinatal death. In this context, this study was planned both to prepare a training programme with evidence of effectiveness and to investigate the effectiveness of perinatal bereavement counselling training for midwives.

DETAILED DESCRIPTION:
The research was planned to be carried out in pretest-posttest control group experimental research design. With the pretest-posttest randomised controlled experimental research method, the effectiveness of the 8-module grief counselling training prepared for women experiencing perinatal grief on the competence of midwives will be examined.

It is planned to carry out 8 modules of bereavement counselling training between December 2024 and December 2025 for midwives actively working in one of the labour, delivery, obstetrics, postpartum, perinatology, septic and aseptic clinics. The study was planned to be carried out with a total of 126 midwives, 63 in the experimental group and 63 in the control group, who responded to the announcement to be made through the social media platforms of associations and organisations to midwives actively working in one of the obstetrics, postpartum, perinatology, septic and aseptic clinics within the borders of Turkey. The link to the web-based scales will be sent to all midwives involved in the study via the WhatsApp programme. The training on perinatal bereavement counselling will be delivered through the Zoom application.

In this trial, randomisation will be used to reduce selection bias in determining the experimental and control groups. A randomisation table from 1 to 126 will be generated using the computerised randomisation programme (https://www.randomizer.org). As the midwives who meet the inclusion criteria are reached, each midwife will be assigned a number and included in the group (experimental or control) with that number. This will determine which participants are in the experimental and control groups.

The planned perinatal bereavement counselling training for midwives will be delivered online and the aim is for midwives to gain skills and competence in perinatal bereavement counselling and to increase their competence in dealing with the problems they may encounter in the counselling process. One group will be the experimental group and the other the control group. In the first part of the study, research brochures will be distributed via social media. These brochures will contain information about the research, the terms and conditions of participation, and contact information for the researchers. In this part, midwives who wish to participate in the research will be contacted via the WhatsApp programme using the research participation brochures distributed on social media platforms. Midwives who wish to participate will be added to the WhatsApp group. One week before the study, the link to the pre-tests will be shared in WhatsApp groups and both groups will be ensured to complete the pre-tests. Participants who do not complete the pre-tests will not be able to participate in the next module. idwives in the experimental group (n = 63) will receive a researcher-developed training on perinatal bereavement counselling for midwives. The training will be reviewed by academics who are experts in their field. The training will be delivered through the online platform ZOOM programme and the training link will be shared in WhatsApp groups before each module. The grief counselling training programme for midwives is as follows:

Module 1: In the first module of the study, midwives who wish to participate in the research will be screened to determine if they meet the inclusion criteria using the research participation brochures distributed through social media platforms. The researcher contact information will be included in the shared brochure and midwives will be able to access the research using this contact information. In order to assess the suitability of midwives who reach the researcher for the study, the initial interview with the midwives will be conducted online via the WhatsApp programme. Midwives who meet the inclusion criteria will be included in the study. Midwives will be randomised into two groups (experimental-control) and separate WhatsApp groups will be created for the two groups. All data collection forms will be created using Google Forms and links to the forms will be sent to participants via these WhatsApp groups. Consent from midwives in both groups will be obtained in some way (verbal or written). Midwives in both groups will be asked to complete pre-tests.

Module 2: Perinatal bereavement counselling training for midwives will be given to midwives in the experimental group who have completed the pre-tests. Module 2 is the introductory part of the training. In the introductory part, general information about the concept of grief is given. This module covers what is grief, what are grief reactions, models of care related to grief, what is perinatal grief (definition, aetiology), psychological characteristics and needs of bereaved families, perinatal grief care in different cultures, models of grief care and communication techniques. The duration of this module is 60 minutes.

Module 3: Midwives who attend the second module will be eligible to attend the third module. The third module consists of two parts. The first part includes training in bereavement counselling for the antenatal period. This part will include the topics of birth preparation, social support and meaning in the prenatal period, birth environment, birth preferences, ensuring privacy and prenatal preparation training. This part should last 60 minutes. The second part is a role play study on counselling women through the trauma process. This part should last 20 minutes.

Module 4: Midwives who participate in the third module can participate in the fourth module. The fourth module includes training in bereavement counselling for the first and second stages of childbirth. In this module, birth pain and non-pharmacological methods of birth pain management will be discussed. This module should last 40 minutes.

Module 5: Midwives who attend the fourth module will be eligible to attend the fifth module. The fifth module consists of two parts. The first part includes training in bereavement counselling for the third and fourth stages of childbirth. This part consists of What does it mean to show the baby the respect it deserves, How it should be, Information support about the baby, Postnatal practices (skin contact, seeing the baby, etc.), Creating memories (photo, hair sample, footprint, blanket, bracelet, etc.), Family support. This part should last 40 minutes. In the second part, work is done on creating memories and role-playing counselling for women in the third and fourth stages of childbirth. This part should last 30 minutes.

Module 6: Midwives who attend the fifth module will be eligible to attend the sixth module. The sixth module consists of two parts. The first part includes training in bereavement counselling for the postpartum period. The first part will cover postpartum care (perineum, wound care, etc.), suppression of lactation, memory storage, the importance of referral when needed, discharge and bereavement education for families, post-discharge bereavement counselling, informing parents for future pregnancies, support for other family members (other children, etc.). This part should last 50 minutes. The second part is a role play study on the provision of postnatal support and counselling. This part should last 20 minutes.

Module 7: Midwives who attend the sixth module will be eligible to attend the seventh module. The seventh module consists of two parts. The first part consists of training midwives to recognise and manage the emotional difficulties they may encounter during the counselling process. This part consists of what is secondary trauma, what are the symptoms of secondary trauma, coping and relaxation techniques and ethical and legal issues in bereavement counselling. This part should last 40 minutes. In the second part, relaxation techniques are practised. This part should last 30 minutes.

Module 8: The last module of the study will be conducted 1 week after the end of the training. Midwives in the experimental group who participated in all modules will be sent a Google Form link for the post-tests via WhatsApp groups. The midwives in the experimental group who completed the post-tests will be asked to complete the training evaluation form in writing in order to evaluate the participation documents. Midwives in the control group will be sent post-tests 1 week after the end of the training process for the experimental group.

Statistical analysis: The data obtained in the research will be analysed using SPSS for Windows (version 22.0, Statistical Package for Social Sciences). Descriptive statistics of continuous variables in the study will be presented with mean and standard deviation values, and descriptive statistics of categorical variables will be presented with frequency and percentage. The distribution of the data will be assessed using the Kolmogorov-Smirnov test and it will be determined that it is suitable for normal distribution. One-way analysis of variance will be used for independent group comparisons, and Tukey post hoc test will be used to identify differences between groups for significant findings. The difference between measurements at different times between the dependent groups was analysed by repeated-measures analysis of variance (repeated-measures ANOVA). In statistical analyses, comparisons with a p-value below 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Midwives who have been active midwives in one of the obstetrics, postnatal, perinatology, septic and aseptic services for at least one year

Exclusion Criteria:

* Academic and freelance midwives
* Midwives who have previously received specialised training in bereavement care

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — women midwives
Enrollment: 126 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Perinatal Bereavement Care Confidence Scale | 1 week before the start of the training and 1 week after the end of the training
  Perinatal Bereavement Care Confidence Scale (PBCCS)The validity and reliability of the scale developed by Kalu et al. in 2019 to evaluate the perinatal grief process and care in this process was developed by Dursun and Akkuş. This measurement tool was developed to determine the grief care confidence of midwives and nurses who provide support to parents experiencing perinatal loss. The scale consists of 35 items and 4 sub-dimensions. The items of the scale, which has a 5-point Likert structure, are scored as strongly agree=5, agree=4, partially agree=3, disagree=2, strongly disagree=1. While the minimum score to be obtained from each dimension is 1, the maximum score is 5. The statements with reversed items are 7, 11 and 33. Low scores obtained from the scale indicate a high level of confidence in perinatal bereavement support. The scale does not have a total score and each factor is scored independently. In the scale; each dimension is evaluated separately within itself.

IPD SHARING:
Plan to Share IPD: No
I donot want to share